CLINICAL TRIAL: NCT01153854
Title: Efficacy, Safety and Cost-effectiveness Analysis of Impact of Racecadotril as an Adjunct in the Treatment of Acute Diarrhea in Mexican Children
Brief Title: Safety, Efficacy and Cost-effectiveness of Racecadotril in Children With Acute Diarrhea in Mexico
Acronym: Raceca-Mex
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Pediatrics, Mexico (Other Government)
Collaborators: Ferrer Laboratories (Unknown)
Responsible Party: Pedro Gutierrez-Castrellon MD, MSc, DSc, National Pediatric Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INP14/2005-Raceca-001
Record Dates: First submitted 2010-06-28; First posted 2010-06-30 (Estimated); Last update posted 2010-06-30 (Estimated); Status verified 2010-06

CONDITIONS: Diarrhea
Keywords: acute diarrhea; Acute diarrhea (three or more watery or semi-watery bowel movements for at least one day lasting no more than 5 days before being admitted)
MeSH Terms: conditions — Diarrhea | interventions — racecadotril

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- ORS-Raceca In hospital Group (Experimental): This group included 135 dehydrated patients which need an oral rehydration therapy in hospital and were assigned to received oral rehydration solution and racecadotril (1.5mg./Kg./t.i.d. doe 5 days) in double blind assigned.
  Interventions: Drug: Racecadotril
- ORS-Placebo in hospital group (Placebo Comparator): This group included 135 dehydrated patients which need an oral rehydration therapy in hospital and were assigned to received oral rehydration solution and placebo in double blind assigned.
  Interventions: Drug: Placebo groups
- ORS-Placebo ambulatory group (Placebo Comparator): This group included 92 non dehydrated patients which were assigned to received oral rehydration solution and placebo in double blind assigned and ambulatory (in home) bases.
  Interventions: Drug: Placebo groups
- ORS-Raceca ambulatory group (Experimental): This group included 92 non dehydrated patients which were assigned to received oral rehydration solution and racecadotril (1.5mg./Kg./t.i.d. doe 5 days) in double blind assigned and ambulatory (in home) bases.
  Interventions: Drug: Racecadotril

INTERVENTIONS:
Drug: Racecadotril — oral racecadotril (1.5mg./Kg./t.i.d. doe 5 days) in double blind assigned.
  Arms: ORS-Raceca In hospital Group; ORS-Raceca ambulatory group
Drug: Placebo groups — Placebo with feature color, appearance and tase similar to racecadotril t.i.d. for 5 days
  Arms: ORS-Placebo ambulatory group; ORS-Placebo in hospital group

SUMMARY:
Rationale: Acute diarrhea (AD) is still a significant morbidity-mortality problem worldwide. Although oral rehydration therapy is the cornerstone, its anti-diarrheal effect is a controversial subject. Since ten years ago, Racecadotrilo´s safety and efficacy had been proved. However, a pharmacoeconomics analysis on this therapeutics has not been published yet.

Objective: Evaluate the efficacy, safety, tolerability and costs associated with Racecadotril administration in comparison to a placebo in infants up to 24 months of age with AD in a hospital (mildly or moderately dehydrated) and ambulatory (no dehydrated) settings at the National Institute of Pediatrics in Mexico.

Material and Methods: Randomized, double-blind, placebo controlled, clinical trial (RDBCCT) with pharmacoeconomics analysis (cost minimization) to realize in 454 infants with AD (270 hospitalized and 184 outpatients), 1 to 24 months of age who concomitantly will receive ORT and Racecadotril (1.5mg./Kg./t.i.d. doe 5 days) (ORT-Rac Group) or placebo (ORT-Placebo Group). The clinical outcomes in the hospitalized infants to measure will be a) Stool output rate at 48hs. and at the end of the study; b) duration of diarrhea; c) percentage of intravenous (IV) needs and d) percentage of adverse events. The outcome variables in outpatient infants to measure will be a) total liquid and semi-liquid bowel movements during the study; b) duration of diarrhea and c) percentage of adverse events. The pharmacoeconomics analysis will involve a cost minimization analysis (CMA). Results will be analyzed through bi and multivariate analysis using STATA 11.0 for Mac, considering a p value < 0.05 as significant. The pharmacoeconomics model will made through decisions trees using TreAge Pro Healthcare v 1.2.0, 2009.

ELIGIBILITY:
Inclusion Criteria:

* children ≥ 1 month of age and ≤ 24 months of age
* Acute diarrhea (defined as three or more watery or semi-watery bowel movements for at least one day lasting no more than 5 days before being admitted)
* For in hospital group: mild or moderate dehydration
* Signed informed consent letter

Exclusion Criteria:

* previous use of oral antibiotics for more than 48 hours (during the two weeks before the trial
* previous use of anti-diarrheal medication (e.g.: bismuth subsalicylate, adsorbents, Loperamide, combinations)
* chronic pathologies (e.g.: cardiopathies, nephropathies, chronic gastrointestinal pathologies, endocrinopathies)

Ages: 1 Month to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 454 (Actual)
Dates: Start 2007-01; Primary Completion 2008-07 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Stool output rate | 2007-2009
  During the study, since the inclusion until the end of the diarrheic episode (24hs after passage of liquid or semiliquid stool) we will measure the stool output rate, reporting it at 48h and at seven day.
Duration of diarrhea | 2007-2009
  In all included patients we will measure the duration of diarrhea, marking as a zero time the moment to sign the informed consent and the end of the diarrheic episod 24hs after the passage of the last liquid or semiliquid stool
Percentage of related adverse events | 2007-2009
  During the duration of the study and five days after we will measure the presence of related adverse events. Any possible event ocurred after sign of consented inform will record and then classified as related or non related and as severe or notr severe adverse event

SECONDARY OUTCOMES:
The pharmacoeconomics analysis | 2007-2009
  The pharmacoeconomics model consisted in a theoretical scheme that makes it possible to conduct simulations of health processes associated with medical care, use of medications, expenses for intravenous hydration and re-hospitalizations secondary to dehydration, through estimates obtained from the efficacy data available from our clinical trial as well as the costs and consequences. The model was prepared using the TreeAge Pro Healthcare v 1.2.0, 2009 software tool

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Gutierrez-Castrellon, MD, MSc, DSc, Principal Investigator — National Pediatric Institute
Locations (1):
- National Pediatric Institute, Mexico City, Mexico City, Mexico

REFERENCES:
- [Background] Szajewska H, Ruszczynski M, Chmielewska A, Wieczorek J. Systematic review: racecadotril in the treatment of acute diarrhoea in children. Aliment Pharmacol Ther. 2007 Sep 15;26(6):807-13. doi: 10.1111/j.1365-2036.2007.03444.x. PMID 17767464
- [Background] Cezard JP, Salazar-Lindo E. Racecadotril in acute diarrhea. Indian Pediatr. 2005 May;42(5):502-3; author reply 503. No abstract available. PMID 15923708
- [Background] Rao SG. Racecadotril (acetorphan) in the treatment of acute watery diarrhoea in children. J Indian Med Assoc. 2002 Aug;100(8):530. No abstract available. PMID 12675192
- [Background] Cojocaru B, Bocquet N, Timsit S, Wille C, Boursiquot C, Marcombes F, Garel D, Sannier N, Cheron G. [Effect of racecadotril in the management of acute diarrhea in infants and children]. Arch Pediatr. 2002 Aug;9(8):774-9. doi: 10.1016/s0929-693x(01)00988-5. French. PMID 12205786
- [Background] Cezard JP, Duhamel JF, Meyer M, Pharaon I, Bellaiche M, Maurage C, Ginies JL, Vaillant JM, Girardet JP, Lamireau T, Poujol A, Morali A, Sarles J, Olives JP, Whately-Smith C, Audrain S, Lecomte JM. Efficacy and tolerability of racecadotril in acute diarrhea in children. Gastroenterology. 2001 Mar;120(4):799-805. doi: 10.1053/gast.2001.22544. PMID 11231932
- [Background] Salazar-Lindo E, Santisteban-Ponce J, Chea-Woo E, Gutierrez M. Racecadotril in the treatment of acute watery diarrhea in children. N Engl J Med. 2000 Aug 17;343(7):463-7. doi: 10.1056/NEJM200008173430703. PMID 10944563